CLINICAL TRIAL: NCT03409367
Title: A Community-based Assessment of Skin Care, Allergies, and Eczema
Acronym: CASCADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Wisconsin, Madison (Other); University of Colorado, Denver (Other); Duke University (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Eric Simpson, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 1R01AR071057-01A1 (NIH); 1R01AR071057-01A1 (NIH)
Record Dates: First submitted 2018-01-11; First posted 2018-01-24 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis; Atopic Disorders; Eczema; Atopic Eczema
Keywords: Prevention; Emollient; Pragmatic clinical trial
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Intervention Model Description: This is a pragmatic, multi-site, randomized community-based trial in which dyads of a parent or legal guardian ("parent") and an infant age 0 to 2 months are enrolled. Participating dyads are randomly assigned to receive lipid-rich emollient with web-based instructions for daily use to infants plus routine skin care instructions (every day moisturizer group) or routine skin care instructions alone (natural skin group). Both groups will receive e-mail and text message reminders to follow protocol instructions based on their group allocation until the infant reaches 24 months old.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, it is not possible blind dyads to the intervention. Administering a placebo emollient is impossible as there are no active ingredients in the emollient and using an emollient that has no barrier improvement properties may irritate the skin. The clinician completing the final assessment will be a blinded assessor.
  Clinic staff will not be informed of participant enrollment or study arm. Parents will be instructed not to disclose their treatment group to clinic staff. Clinicians and clinic staff will direct participants to follow skin care recommendations as described by the study materials.
  Blinded researchers will be responsible for health record review to collect the primary outcome. At completion of health record review, researchers will complete a form measuring whether the assessor became unblinded while reviewing the record.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Emollient (Experimental): Parent-infant dyads assigned to the intervention arm receive a lipid-rich emollient and educational materials promoting once daily full-body emollient use until the infant is 24 months old. Parents select one of five emollients to be mailed to the dyad's home at enrollment and approximately every six months for the duration of the study. These emollients include (1) CeraVe Healing Ointment, (2) Vaseline, (3) Cetaphil cream, (4) CeraVe cream, and (5) Vanicream.
  Interventions: Other: Participant choice of over-the-counter emollients: Vaseline, Vanicream, CeraVe Healing Ointment, CeraVe cream, Cetaphil cream
- Natural Skin (No Intervention): Parent-infant dyads assigned to the control arm receive educational materials promoting general infant skin care guidelines only and are asked to refrain from emollient use unless dry skin develops (current standard of care guidelines).

INTERVENTIONS:
Other: Participant choice of over-the-counter emollients: Vaseline, Vanicream, CeraVe Healing Ointment, CeraVe cream, Cetaphil cream — Lipid-rich emollient serving as skin barrier
  Arms: Daily Emollient

SUMMARY:
Atopic dermatitis (AD) affects over 9 million children in the U.S. and often heralds the development of asthma, food allergy, skin infections and neurodevelopmental disorders. Recent advances identify skin barrier dysfunction to be the key initiator of AD and possibly allergic sensitization.

Our central hypothesis is that daily emollient use from birth can prevent the development of AD in a community setting and into newborns unselected for risk. The results of a community-based clinical trial utilizing a pragmatic trial design will be immediately applicable to the population at large and will establish a new standard of care for all newborns.

DETAILED DESCRIPTION:
AD affects over 9 million children in the U.S. and ranks first among all skin conditions in global disability burden. AD often heralds the development of several comorbidities including asthma, food allergy, skin infections and neurodevelopmental disorders. Because of the significant socioeconomic impact of atopic dermatitis and its effect on the quality of life of children and families, there have been decades of research focused on prevention with limited success. Recent advances in cutaneous biology identify epidermal defects and skin barrier dysfunction to be the key initiators of atopic dermatitis and possibly allergic sensitization. Our central hypothesis is that emollient therapy from birth can prevent the development of AD. The findings of this trial will support the development of evidence-based skin care clinical guidelines for infants that currently do not exist. Recently, our international multi-centered clinical trial found enhancing early skin barrier function with daily emollient use from birth significantly reduces the risk of AD development in high-risk populations by 50%. With CASCADE, we extend this work into the community setting and into newborns unselected for risk, so results will be immediately applicable to the population at large and will establish a new standard of care for all newborns.

The specific aims are as follows:

1. Perform a community-based pragmatic randomized controlled trial investigating whether daily full-body emollient application starting in the first 2 months of life prevents atopic dermatitis in a real-world setting. The population for this trial consists of newborns between 0-2monthsof age, not selected for risk. Recruitment of families will occur during the course of routine care within primary care offices that are members of practice-based research networks(PBRNs).The intervention includes general skin care recommendations plus full-body daily lipid-rich emollient use. The control population will receive general skin care advice only and refrain from daily emollient use. The primary outcome will be the cumulative incidence of atopic dermatitis at age 24 months as determined by blinded clinicians trained in the diagnosis of AD. Key secondary clinical outcomes include time to disease onset and incidence of self-reported food allergy and wheeze using parental questionnaires.
2. As an exploratory aim, determine whether a family history of allergic disease and key early life exposures such as pet ownership modify the preventive effect of emollient therapy on atopic dermatitis. While the primary objective of this clinical trial is to determine the effectiveness of an emollient intervention in a real-world setting, data will be gathered on allergy history in the family and pet ownership-variables that may modify the effect of emollient therapy. Future implementation studies may target subpopulations found most likely to benefit from emollient intervention.

Twenty-five primary care clinics that participate in PBRNs from Oregon, Colorado, Wisconsin and North Carolina are the setting for the study protocol. The expected results from this project would represent a major public health breakthrough with the potential for reducing the atopic disease burden on a global scale.

ELIGIBILITY:
Inclusion Criteria:

* Parent can provide electronic signed and dated informed consent form.
* Parent is willing and able to comply with all study procedures for the duration of the study.
* Parent is a primary caretaker of an infant 0 to 2 months of age.
* Parent is 18 years of age or older at time of consent.
* Parent can speak, read, and write in English or Spanish.
* Parent has a valid e-mail address or phone that can receive text messages
* Parent has reliable access to the internet.
* Infant is a patient of a participating Meta-LARC clinic site at the time of consent.

Exclusion Criteria:

* Infant was born at less than 25 weeks gestational age.
* Infant has established eczema as diagnosed by the primary healthcare provider at clinic site of enrollment per parent report.
* Infant has known adverse reaction to petrolatum-based emollients.
* Infant has an immunodeficiency genetic syndrome such as Wiskott-Aldrich Syndrome or Severe Combined Immunodeficiency Syndrome.
* Infant has extremely low birth weight (less than 1000g or 2.2 lbs at birth).
* Infant has a sibling enrolled in the study.
* Parent is unwilling or unable to comply with study procedures.

Ages: 1 Day to 63 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1260 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Simpson, MD, Principal Investigator — Oregon Health and Science University
Locations (4):
- United States (4):
  - University of Colorado-Denver, Denver, Colorado
  - Duke University, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be according to the NIAMS guidelines
Supporting Information: Study Protocol, SAP
Time Frame: Supporting information will be shared per NIAMS guidelines

REFERENCES:
- [Derived] Simpson EL, Michaels LC, Ramsey K, Fagnan LJ, Nease DE, Henningfield M, Dolor RJ, Lapidus J, Martinez-Ziegenfuss X, Vu A, Ferrara L, Zuckerman KE, Morris CD, Williams HC; CASCADE Consortium. Emollients to Prevent Pediatric Eczema: A Randomized Clinical Trial. JAMA Dermatol. 2025 Jul 23;161(9):957-65. doi: 10.1001/jamadermatol.2025.2357. Online ahead of print. PMID 40699587
- [Derived] Eichner B, Michaels LAC, Branca K, Ramsey K, Mitchell J, Morris CD, Fagnan LJ, Dolor RJ, Elder N, Hahn DL, Nease DE, Lapidus J, Cibotti R, Block J, Simpson EL. A Community-based Assessment of Skin Care, Allergies, and Eczema (CASCADE): an atopic dermatitis primary prevention study using emollients-protocol for a randomized controlled trial. Trials. 2020 Mar 4;21(1):243. doi: 10.1186/s13063-020-4150-5. PMID 32131885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from 25 community-based primary care sites in four states (Oregon, North Carolina, Wisconsin, Colorado) from July 2018-February 2021.
Groups:
- Daily Emollient: Parents assigned to the intervention arm receive a lipid-rich emollient and educational materials promoting once daily full-body emollient use until infant age 24 months. Participant choice of over-the-counter emollients: Vaseline, Vanicream, CeraVe Healing Ointment, CeraVe cream, Cetaphil cream: Lipid-rich emollient serving as skin barrier
- Natural Skin: Parents assigned to the control arm receive educational materials promoting general infant skin care guidelines only and asked to refrain from emollient use unless dry skin develops (current standard of care guidelines).
Period: Overall Study
Arm/Group | Daily Emollient | Natural Skin
Started | 623 | 637
Enrolled Infants | 623 | 637
Enrolled Parents (At least 623 parents were enrolled in the "Daily Emollient" Arm/Group and at least 637 parents were enrolled in the "Natural Skin" Arm/Group, however, it is unknown how many total parents were enrolled for each of the Arms/Groups. A single parent or guardian gave consent for dyad participation. Each dyad involves an infant and a parent.) | 623 | 637
Completed | 603 | 625
Not Completed | 20 | 12

BASELINE CHARACTERISTICS:
Population: Parent-infant dyads contributing sufficient survey or chart data to be included in the intent-to-treat analysis. All data collected and reported relates to information about the infant. No baseline or follow-up data is collected about parents.
Groups:
- Natural Skin: Parents assigned to the control arm receive educational materials promoting general infant skin care guidelines only and to refrain from emollient use unless dry skin develops (current standard of care guidelines).
- Total: Total of all reporting groups
Arm/Group | Daily Emollient | Natural Skin | Total
Number analyzed (Participants) | 603 | 625 | 1228
Age, Continuous [Mean (Standard Deviation); unit: Days] | 23.9 (16.0) | 24.0 (16.6) | 23.9 (16.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 324 | 350 | 674
  Female | 279 | 274 | 553
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 144 | 141 | 285
  Not Hispanic or Latino | 437 | 459 | 896
  Unknown or Not Reported | 22 | 25 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 2 | 15
  Asian | 19 | 16 | 35
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 44 | 41 | 85
  White | 439 | 473 | 912
  More than one race | 59 | 53 | 112
  Unknown or Not Reported | 27 | 38 | 65

OUTCOME MEASURES:

1. Primary Outcome: Provider-diagnosed Atopic Dermatitis
Description: The cumulative incidence of AD as recorded in health records. Trained clinicians will assess for AD at each clinic visit and record in the health record.
Time Frame: up to 24 months
Population: Diagnosis of atopic dermatitis recorded by primary care clinicians in health records by 24 (+/- 3) months of age. Multiple imputation of 199 missing outcomes (92 intervention, 107 control). All ITT with multiple imputation for participants with absent outcome data. Numbers represent participants per randomized arm, regardless of adherence to instructions. Counts were summarized over 15 multiple imputation datasets generated by chained equations using baseline and follow-up survey responses.
Measure: Number; unit: Participants with imputed values
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 603 | 625
Participants with imputed values | 217.7 | 268.5
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the cumulative incidence of atopic dermatitis does not differ between the Daily Emollient and Natural Skin arms, or that the risk ratio is equal to 1; Test type: Equivalence — The risk ratio is equal to 1; p = 0.019, Regression, log-binomial; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.73 to 0.97] — Adjusted for family history of atopy (stratified randomization) and primary care site. Adjusted for multiple imputations

2. Secondary Outcome: Parent Report of Atopic Dermatitis
Description: Parent or guardian reports that a clinician has diagnosed their child with atopic dermatitis (eczema) at any quarterly contact up to 24 months of age.
Time Frame: up to 24 months
Population: Multiple imputation of 111 outcomes considered missing when parent did not respond at 21 or 24 months and no diagnosis had been reported at earlier contacts. All ITT with multiple imputation for 9% of participants with absent outcome data. Numbers represent participants according to arm randomized, regardless of adherence to study instructions. Counts were summarized over 15 multiple imputation datasets generated by chained equations using baseline and follow-up survey responses.
Measure: Number; unit: Participants with imputed values
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 603 | 625
Participants with imputed values | 161.1 | 219.1
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the cumulative incidence of parent-reported AD does not differ between the Daily Emollient and Natural Skin arms, or that the risk ratio (RR) is equal to 1; Test type: Equivalence — The risk ratio (RR) is equal to 1; p = 0.002, Regression, log-binomial; Adjusted for family history of atopy (stratified randomization) and primary care site. Adjusted for multiple imputations; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.65 to 0.90]

3. Secondary Outcome: Atopic Dermatitis by UK Working Party Criteria
Description: Parental report of AD using UK Working Party criteria. Parent responds "yes" to all parts of a modified version of the UK Working Party criteria at 12 and/or 24 month. Criteria include an itchy rash in flexural areas, generally dry skin, and asthma or hay fever in a first-degree relative.
Time Frame: up to 24 months
Population: Multiple imputation of 148 outcomes considered missing when parent did not respond at 24 months and the previous 12-month contact was not positive for AD by these criteria. All ITT with multiple imputation for 12% of participants with absent outcome data. Numbers represent participants according to arm randomized, regardless of adherence to study instructions. Counts were summarized over 15 multiple imputation datasets generated by chained equations using baseline and follow-up survey responses.
Measure: Number; unit: Participants with imputed values
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 603 | 625
Participants with imputed values | 72.3 | 83.1
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the cumulative incidence of AD by modified UK Working Party criteria does not differ between the Daily Emollient and Natural Skin arms, or that the risk ratio (RR) is equal to 1; Test type: Equivalence — Risk ratio is equal to 1; p = 0.323, Regression, log-binomial — Adjusted for family history of atopy (stratified randomization) and primary care site. Adjusted for multiple imputations; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.65 to 1.15]

4. Secondary Outcome: Atopic Dermatitis by Children's Eczema Questionnaire
Description: AD as diagnosed by the Children's Eczema Questionnaire (CEQ). Parent response to 3 CEQ questions is consistent with AD at 12 and/or 24 months of age.
Time Frame: up to 24 months
Population: Multiple imputation of 136 outcomes considered missing when parent did not respond at 24 months and the previous 12-month contact was not positive for AD by these criteria. All ITT with multiple imputation for 11% of participants with absent outcome data. Numbers represent participants according to arm randomized, regardless of adherence to study instructions. Counts were summarized over 15 multiple imputation datasets generated by chained equations using baseline and follow-up survey responses.
Measure: Number; unit: Participants with imputed values
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 603 | 625
Participants with imputed values | 156.9 | 195.3
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the cumulative incidence of AD by CEQ does not differ between the Daily Emollient and Natural Skin arms, or that the risk ratio (RR) is equal to 1; Test type: Equivalence — Risk ratio is equal to 1; p = 0.044, Regression, log-binomial; [statistical method as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.70 to 0.99]

5. Secondary Outcome: Atopic Dermatitis With Prescription or Over-the-counter Therapies in Chart
Description: Cumulative incidence of provider-diagnosed AD requiring prescription or over-the-counter therapies from chart review. Health records at primary care practice includes both a diagnosis of AD and prescription and/or over-the-counter (OTC) therapies. Prescription therapies could be steroids, calcineurin inhibitors, crisaborole, or antibacterials. OTC therapies could be steroids or antihistamines.
Time Frame: up to 24 months
Population: Multiple imputation of 199 missing outcomes. All ITT with multiple imputation for 16% of participants with absent outcome data. Numbers represent participants according to arm randomized, regardless of adherence to study instructions. Counts were summarized over 15 multiple imputation datasets generated by chained equations using baseline and follow-up survey responses.
Measure: Number; unit: Participants with imputed values
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 603 | 625
Participants with imputed values | 116.5 | 179.8
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the cumulative incidence of AD with prescription or OTC therapies in the health record does not differ between the Daily Emollient and Natural Skin arms, or that the risk ratio (RR) is equal to 1; Test type: Equivalence — The risk ratio (RR) is equal to 1; p = 0.0004, Regression, log-binomial; [statistical method as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.68, 95% CI 2-sided [0.55 to 0.84]

6. Secondary Outcome: Atopic Dermatitis With or Without Prescription or Over-the-counter Therapies in Chart (Ordinal)
Description: Ordinal coding of diagnosis of atopic dermatitis (eczema) in primary care health records, coded as none, eczema without prescription or over-the-counter (OTC) topical therapies, eczema with OTC only, or eczema with prescription therapies. Prescription therapies could be steroids, calcineurin inhibitors, crisaborole, or antibacterials. OTC therapies could be steroids or antihistamines.
Time Frame: Up to 24 months
Population: All ITT with multiple imputation for 16% of participants with absent outcome data. Numbers represent participants according to arm randomized, regardless of adherence to study instructions. Counts were summarized over 15 multiple imputation datasets generated by chained equations using baseline and follow-up survey responses.
Measure: Number; unit: Participants with imputed values
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 603 | 625
Participants with imputed values
  No atopic dermatitis | 385.3 | 356.5
  Atopic dermatitis without topical medication | 101.2 | 88.7
  Atopic dermatitis with over-the-counter therapy | 38.3 | 59.7
  Atopic dermatitis with prescription therapy | 78.2 | 120.1
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the odds of belonging to the next higher category of severity are equal in the Daily Emollient and Natural Skin arms; Test type: Equivalence — The odds ratio (OR) is equal to 1. An OR < 1 could be considered evidence that daily emollient use is associated with lower severity of AD, as operationalized here by the type of recommended treatment; p = 0.004, Regression, proportional odds — Adjusted for family history of atopy (stratified randomization) and primary care site. Adjusted for multiple imputations of 199 missing outcomes; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.55 to 0.89]

7. Secondary Outcome: Prescribed or Over-the-counter Topical Skin Medication by Parent Report
Description: Ordinal formulation of parent report: no AD, AD not treated with steroidal or non-steroidal cream or ointment ("therapy"), AD treated with over-the-counter (OTC) therapy, AD treated with prescription therapy. AD could be reported on annual questionnaires or quarterly contacts. Therapies reported on annual questionnaires.
Time Frame: up to 24 months
Population: Participants with (a) a parent report of provider diagnosis from an annual questionnaire or quarterly contact or (b) if no diagnosis, a parent response to a quarterly or annual contact at 21 to 24 months. Numbers represent participants according to arm randomized, regardless of adherence to study instructions.
Measure: Number; unit: participants
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 561 | 556
participants
  No AD | 410 | 364
  AD, no topical OTC or Rx reported | 36 | 52
  OTC topical | 31 | 38
  Rx and/or OTC topical | 84 | 102
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; [analysis description as in outcome 6, analysis 1]; Test type: Equivalence — Odds ratio (OR) is equal to 1. An OR < 1 could be considered evidence that daily emollient use is associated with lower severity of AD, as operationalized here by the type of treatment; p = 0.013, Regression, proportional odds; Adjusted for family history of atopy (stratified randomization) and primary care site; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.56 to 0.93]

8. Secondary Outcome: Skin Infections Diagnosed and Recorded in Chart Review
Description: Chart outcome for provider diagnosis or medications associated with skin infections, including topical antibiotics. Skin infection diagnoses include impetigo, candida, wart/verruca, molluscum, or herpes simplex.
Time Frame: up to 24 months
Population: All participants with (a) at least one primary care visit between 20 and 27 months of age or (b) a skin infection diagnosis earlier than 20 months. Numbers represent participants according to arm randomized, regardless of adherence to study instructions.
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 509 | 506
Participants | 101 | 107
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the cumulative incidence of skin infections in the health record does not differ between the Daily Emollient and Natural Skin arms; Test type: Equivalence — The risk ratio (RR) is equal to 1; p = 0.509, Regression, log-binomial; Adjusted for family history of atopy (stratified randomization) and primary care site; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.73 to 1.17]

9. Secondary Outcome: Provider-diagnosed Asthma
Description: Health records at primary care practice include at least one diagnosis of asthma.
Time Frame: up to 24 months
Population: All participants with (a) at least one primary care visit between 20 and 27 months of age or (b) asthma diagnosis earlier than 20 months. Numbers represent participants according to arm randomized, regardless of adherence to study instructions.
Measure: Number; unit: participants
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 503 | 494
participants | 14 | 13
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the cumulative incidence of asthma in the health record does not differ between the Daily Emollient and Natural Skin arms, or that the risk ratio (RR) is equal to 1; Test type: Equivalence — The risk ratio is equal to 1; p = 0.900, Regression, log-binomial; Adjusted for family history of atopy (stratified randomization) and primary care site; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.50 to 2.18]

10. Secondary Outcome: Severity of AD Symptoms Using POEM
Description: Patient-Oriented Eczema Measure (POEM) score, elicited from families of infants who reported AD diagnosis at this or any previous contact or whose CEQ response indicated AD. The POEM has seven items and ranges from 0 to 28, with higher scores reflecting more severe symptoms of AD.
Time Frame: 12 months of age
Population: Respondents to 12-month questionnaires who reported a provider diagnosis of AD in the same questionnaire or at a quarterly contact, or whose response to the CEQ indicated AD. Numbers represent participants according to arm randomized, regardless of adherence to study instructions.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 128 | 165
score on a scale | 3 [1 to 7] | 2 [0 to 5]
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the odds of belonging to the next higher category of severity are equal in the Daily Emollient and Natural Skin arms, or that the ordinal odds ratio (OR) is equal to 1; Test type: Equivalence — An ordinal OR < 1 could be considered evidence that daily emollient use is associated with lower severity of AD symptoms among those diagnosed with AD; p = 0.064, Regression, proportional odds; Adjusted for family history of atopy (stratified randomization); Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.98 to 2.21] — The daily emollient is in the numerator and the natural skin is in the denominator

11. Secondary Outcome: Severity of AD Symptoms Using POEM
Description: as for outcome 10
Time Frame: 24 months of age
Population: Respondents to 24-month questionnaires who reported a provider diagnosis of AD in the same or previous annual questionnaire or at a quarterly contact, or whose response to the CEQ indicated AD. Numbers represent participants according to arm randomized, regardless of adherence to study instructions.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 185 | 216
score on a scale | 2 [0 to 5] | 1 [0 to 4]
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; [analysis description as in outcome 10, analysis 1]; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p = 0.007, Regression, proportional odds; Adjusted for family history of atopy (stratified randomization); Odds Ratio (OR) = 1.62, 95% CI 2-sided [1.14 to 2.30] — Daily emollient in the numerator and natural skin in the denominator

12. Secondary Outcome: Severity of AD Symptoms Using IDQoL
Description: Symptom severity as reflected by the Infant Dermatology Quality of Life Instrument (IDQoL) elicited from families of infants who reported AD diagnosis at this or any previous contact or whose CEQ response indicated AD. The IDQoL has 12 items and ranges from 0-37 with higher scores reflecting greater adverse effect of AD on quality of life
Time Frame: 12 months
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 128 | 165
score on a scale | 4 [2 to 7] | 4 [1 to 6]
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; [analysis description as in outcome 10, analysis 1]; Test type: Equivalence — The ordinal odds ratio (OR) is equal to 1. An OR < 1 could be considered evidence that daily emollient use is associated with lower severity of AD symptoms among those diagnosed with AD; p = 0.070, Regression, proportional odds; Adjusted for family history of atopy (stratified randomization); Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.97 to 2.18] — Daily moisturizer is the numerator and natural skin is the denominator

13. Secondary Outcome: Severity of AD Symptoms Using IDQoL
Description: as for outcome 12
Time Frame: 24 months
Population: Respondents to 24-month questionnaires who reported a provider diagnosis of AD in the same questionnaire or at a quarterly contact, or whose response to the CEQ indicated AD. Numbers represent participants according to arm randomized, regardless of adherence to study instructions.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 184 | 216
score on a scale | 3 [1.5 to 6] | 3 [1 to 5]
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the odds of belonging to the next higher category of severity are equal in the Daily Emollient and Natural Skin arms, or that the odds ratio (OR) is equal to 1. An OR < 1 could be considered evidence that daily emollient use is associated with lower severity of AD symptoms among those diagnosed with AD; Test type: Equivalence — Odds ratio (OR) is equal to 1. An OR < 1 could be considered evidence that daily emollient use is associated with lower severity of AD symptoms among those diagnosed with AD; p = 0.085, Regression, proportional odds; Adjusted for family history of atopy (stratified randomization); Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.96 to 1.91]

14. Secondary Outcome: Food Allergy Symptoms
Description: Parent reports immediate food allergy reaction in child at 12- or 24-month questionnaire, or both.
Time Frame: 12 months, 24 months or both
Population: Respondents who answered items about immediate food allergy symptoms. Numbers represent participants according to arm randomized, regardless of adherence to study instructions.
Measure: Number; unit: participants
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 549 | 544
participants | 59 | 77
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the cumulative incidence of immediate food allergy reactions does not differ between the Daily Emollient and Natural Skin arms, or that the risk ratio (RR) is equal to 1; Test type: Equivalence — The risk ratio (RR) is equal to 1; p = 0.079, Regression, log-binomial; Adjusted for family history of atopy (stratified randomization) and primary care site; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.55 to 1.03]

15. Secondary Outcome: Food Allergy Diagnosis With Positive Test
Description: Parent reports a provider diagnosis of and a positive test for food allergy at 12- or 24-month questionnaire, or both.
Time Frame: up to 24 months
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 550 | 548
participants | 16 | 18
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the cumulative incidence of food allergies does not differ between the Daily Emollient and Natural Skin arms, or that the risk ratio (RR) is equal to 1; Test type: Equivalence — Risk ratio (RR) is equal to 1; p = 0.669, Regression, log-binomial; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.45 to 1.66]

16. Secondary Outcome: Primary Outcome of Provider-diagnosed Atopic Dermatitis
Description: Diagnosis of atopic dermatitis (eczema) recorded by primary care providers in health records up to 12 months of age (rather than 24 months).
Time Frame: up to 12 months
Population: Infants with diagnosis of atopic dermatitis at <=12 months or with no diagnosis and at least one primary care visit in the health record after 9 months of age. Numbers represent participants according to arm randomized, regardless of adherence to study instructions.
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 586 | 589
Participants | 115 | 151
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the cumulative incidence of AD does not differ between the Daily Emollient and Natural Skin arms, or that the risk ratio (RR) is equal to 1. Alternatively, a RR < 1 could be considered evidence that daily emollient is associated with lower incidence of AD; Test type: Equivalence — Risk ratio (RR) is equal to 1. Alternatively, a RR < 1 could be considered evidence that daily emollient is associated with lower incidence of AD; p = 0.013, Regression, log-binomial; Adjusted for family history of atopy (stratified randomization) and primary care site; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.62 to 0.95]

17. Secondary Outcome: Provider-diagnosed Atopic Dermatitis at 18 Months
Description: Diagnosis of atopic dermatitis (eczema) recorded by primary care providers in health records up to 18 months of age.
Time Frame: up to 18 months
Population: Infants with diagnosis of atopic dermatitis at <=18 months or with no diagnosis and at least one primary care visit in the health record after 15 months of age. Numbers represent participants according to arm randomized, regardless of adherence to study instructions.
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 561 | 570
Participants | 154 | 196
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; [analysis description as in outcome 16, analysis 1]; Test type: Equivalence — [test comment as in outcome 16, analysis 1]; p = 0.009, Regression, log-binomial; Adjusted for family history of atopy (stratified randomization) and primary care site; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.67 to 0.94]

18. Other Pre Specified Outcome: Provider-diagnosed Atopic Dermatitis - Low-risk Population
Description: Subgroup population: In the subgroup of participants who did not report atopic dermatitis in a first-degree relative, diagnosis of atopic dermatitis (eczema) recorded by primary care providers in health records
Time Frame: up to 24 months
Population: All ITT with multiple imputation for 19% of participants with absent outcome data. Numbers represent participants according to arm randomized, regardless of adherence to study instructions. Counts were summarized over 15 multiple imputation datasets generated by chained equations using baseline and follow-up survey responses.
Measure: Number; unit: Participants with imputed values
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 307 | 322
Participants with imputed values | 102.1 | 139.7
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; The null hypothesis is that the cumulative incidence of AD does not differ between the Daily Emollient and Natural Skin arms, or that the risk ratio (RR) is equal to 1; Test type: Equivalence — Risk ratio (RR) is equal to 1; p = 0.012, Regression, log-binomial; Adjusted for primary care site. Adjusted for multiple imputations of 121 missing outcomes; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.63 to 0.94]

19. Other Pre Specified Outcome: Provider-diagnosed Atopic Dermatitis - High-risk Population
Description: Subgroup population: In the subgroup of participants who reported atopic dermatitis in a first-degree relative, diagnosis of atopic dermatitis (eczema) recorded by primary care providers in health records
Time Frame: up to 24 months
Population: All ITT with multiple imputation for 13% of participants with absent outcome data. Numbers represent participants according to arm randomized, regardless of adherence to study instructions. Counts were summarized over 15 multiple imputation datasets generated by chained equations using baseline and follow-up survey responses.
Measure: Number; unit: Participants with imputed values
Arm/Group | Daily Emollient | Natural Skin
Number analyzed (Participants) | 296 | 303
Participants with imputed values | 115.7 | 128.7
Statistical Analysis 1: Comparison: Daily Emollient vs Natural Skin; [analysis description as in outcome 18, analysis 1]; Test type: Equivalence — Risk ratio (RR) is equal to 1; p = 0.303, Regression, log-binomial; Adjusted for primary care site. Adjusted for multiple imputations of 78 missing outcomes; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.73 to 1.10]

ADVERSE EVENTS:
Time Frame: 2 years (enrollment through 24 months +/- 3 months)
Description: Serious adverse events = hospitalization and new major medical condition Adverse events = reaction to a skincare product All-Cause Mortality Population included = Infants only. Serious adverse events, adverse events and all-cause mortality were not monitored/assessed for parents.
  All recorded events reported by participants or identified on chart audit.
Groups:
- Daily Emollient: Daily Emollients: Infants assigned to the intervention arm receive a lipid-rich emollient and educational materials promoting once daily full-body emollient use until infant age 24 months. Participant choice of over-the-counter emollients: Vaseline, Vanicream, CeraVe Healing Ointment, CeraVe cream, Cetaphil cream: Lipid-rich emollient serving as skin barrier.
- Natural Skin: Natural Skin: Infants assigned to the control arm receive educational materials promoting general infant skin care guidelines only and asked to refrain from emollient use unless dry skin develops (current standard of care guidelines).
Arm/Group | Daily Emollient | Natural Skin
All-Cause Mortality (participants affected / at risk) | 1/614 | 1/633
Serious Adverse Events (participants affected / at risk) | 25/614 | 39/633
Other Adverse Events (participants affected / at risk) | 134/614 | 155/633
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Emollient (N=614) | Natural Skin (N=633)
Acute leukemia, acute myeloid leukemia NOS, eosinophilic pustular folliculitis (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Laryngomalacia, Kabuki make-up syndrome, macrocephaly (Congenital, familial and genetic disorders) | 1 (1) | 2 (2)
Gastritis acute, gastroenteritis, gastrointestinal disorder NOS, oropharyngeal dysphagia, vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5)
Intussusception, inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Periodic Fever Syndrome (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Milk allergy (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis viral, COVID-19, influenza, pneumonia, rhinovirus NOS, thrush, viral infection (Infections and infestations) | 4 (4) | 6 (6)
Asphyxia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chemical burn of esophagus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture NOS, subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Dehydration, failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Sagittal craniosynostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Choledochal cyst, neuroblastoma, Langerhans cell histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Autism spectrum disorder (Nervous system disorders) | 1 (1) | 3 (3)
Brain empyema, epilepsy NOS, episodic ataxia, febrile seizure, neonatal seizure disorder (Nervous system disorders) | 3 (3) | 4 (4)
Meningitis bacterial (Nervous system disorders) | 0 (0) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Breath holding spells, bronchial hyper-reactivity, bronchiolitis, croup infectious, RSV, URI (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 16 (17)
Cleft palate repair, Nissen fundoplication (Surgical and medical procedures) | 1 (1) | 1 (1)
Subgaleal haemorrhage (Vascular disorders) | 0 (0) | 1 (2)
Hospitalization (Investigations) | 1 (1) | 0 (0) — Hospitalization reported, no further information available
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Emollient (N=614) | Natural Skin (N=633)
Eosinophilic pustular folliculitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Allergic reaction NOS, urticaria (Immune system disorders) | 2 (2) | 4 (4)
Acne infantile (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 30 (35) | 40 (46)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (8) | 7 (8)
Eczema (Skin and subcutaneous tissue disorders) | 22 (26) | 26 (38)
Eczema exacerbated (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 89 (122) | 99 (127)
Scarlet fever (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin infection / Staphylococcal skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin sensitization (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Viral rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT03409367/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT03409367/SAP_001.pdf